CLINICAL TRIAL: NCT01336140
Title: Attenuation of the Side Effect Profile Of Regadenoson: A Randomized Double-Blind Placebo-Controlled Study With Aminophylline in Patients Undergoing Myocardial Perfusion Imaging and Have Severe Chronic Kidney Disease (ASSUAGE-CKD Trial)
Brief Title: Attenuation of the Side Effect Profile of Regadenoson: Study With Aminophylline in Patients With Severe Kidney Disease Undergoing Myocardial Perfusion Imaging
Acronym: ASSUAGE-CKD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Rami Doukky, Director of Nuclear Cardiology and Stress Testing Laboratories, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ASSUAGE-CKD; 110129 (Other: FDA - IND)
Record Dates: First submitted 2011-04-11; First posted 2011-04-15 (Estimated); Results first posted 2013-02-13 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Patients With Severe Chronic Kidney Disease Being Evaluated With Nuclear Stress Testing of the Heart Using the Stress Agent Regadenoson
Keywords: regadenoson; chronic kidney disease; renal failure; lexiscan; aminophylline; SPECT; Myocardial Perfusion Imaging; pharmacologic stress test; Patients with stage IV or V chronic kidney disease being assessed with nuclear stress testing of the heart using the stress agent regadenoson (Lexiscan ®)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency | interventions — Aminophylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aminophylline (Experimental): 75 mg of intravenous aminophylline.
  Interventions: Drug: Aminophylline
- Placebo (Placebo Comparator): Matching 0.9 Normal Saline (sterile salt water)administered intravenously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aminophylline — 75 mg of intravenous aminophylline
  Arms: Aminophylline
Drug: Placebo — Matching 0.9 Normal Saline (sterile salt water)administered intravenously.
  Arms: Placebo

SUMMARY:
The routine administration of 75 mg of intravenous aminophylline in patients with severe chronic kidney disease undergoing a nuclear stress test with regadenoson (Lexiscan®) can reduce or eliminate the incidence of diarrhea and other side effects related to regadenoson.

DETAILED DESCRIPTION:
Approximately 300 patients with severe chronic kidney disease who are referred for a nuclear stress testing of the heart with regadenoson (Lexiscan®) will be recruited to participate in the study. Following regadenoson (administered as part of a stress routine test protocol) participants will receive either aminophylline (75 mg - intravenously) or a matching inactive placebo (sterile salt water) injection. Participants will be surveyed for gastrointestinal symptoms and other side effects related to regadenoson. The frequency and severity of such side effects will be compared between the two study groups (aminophylline vs. placebo).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients referred to undergo a clinically-indicated regadenoson-stress myocardial perfusion imaging at Rush University Medical Center
* Stage IV or V chronic kidney disease (GFR < 30, hemodialysis, and/or peritoneal dialysis).

Exclusion Criteria:

* Patient refusal to participate
* Known allergic reaction to aminophylline.
* Pre-existing headache or acute/subacute GI illness with symptoms of diarrhea, abdominal discomfort, nausea or vomiting.
* Any contraindication to aminophylline: hypotension, unstable cardiac arrhythmias and acute coronary symptoms.
* Uncontrolled seizure disorder defined as more than 2 seizure episodes in the past 12 months or any seizure in the past week.
* Pregnant or breast-feeding women.
* Patients receiving anti-platelet agent dipyridamole (Persantine® or Aggrenox®).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rami Doukky, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Doukky R, Rangel MO, Dick R, Wassouf M, Alqaid A, Margeta B. Attenuation of the side effect profile of regadenoson: a randomized double-blind placebo-controlled study with aminophylline in patients undergoing myocardial perfusion imaging and have severe chronic kidney disease--the ASSUAGE-CKD trial. Int J Cardiovasc Imaging. 2013 Jun;29(5):1029-37. doi: 10.1007/s10554-012-0166-6. Epub 2012 Dec 11. PMID 23224354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the period from June 14, 2011 to May 14, 2012 in the stress testing laboratories of Rush University medical center and John H. Stroger, Jr. Hospital of Cook County (Chicago, IL.
Pre-assignment Details: 427 patients were recruited. 122 patients were excluded: 50 refused; 35 met an exclusion criteria; 1 was previously enrolled in the trial; 26 had a contraindication to aminophylline. 5 consenting subjects were excluded: 3 had their regadenoson-stress clinically cancelled; 2 treatment assignment could not be verified (labeling error).
Period: Overall Study
Arm/Group | Aminophylline | Placebo
Started | 150 | 150
Completed | 150 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aminophylline | Placebo | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 125 | 111 | 236
  >=65 years | 25 | 39 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (13) | 56 (13) | 55 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 54 | 107
  Male | 97 | 96 | 193
Region of Enrollment [Number; unit: participants]
  United States | 150 | 150 | 300

OUTCOME MEASURES:

1. Primary Outcome: Diarrhea (as Reported by the Patient)
Description: Number of patients who report any incident of diarrhea. Patients will be surveyed for incidents of diarrhea following to the completion of the cardiac stress testing procedure and prior to discharge from the laboratory (typically within 2 hours from stress completion).
  The primary endpoint encompasses the number of patients with reported symptoms of diarrhea, not the number of bowel movements.
Time Frame: Within 2 hours from the intervention
Population: All patients.
Measure: Number; unit: participants
Arm/Group | Aminophylline | Placebo
Number analyzed (Participants) | 150 | 150
participants | 9 | 26
Statistical Analysis 1: Comparison: Aminophylline vs Placebo; We calculated that a minimum of 248 subjects are needed to attain 80% power to detect 70% reduction in the incidence of the primary endpoint (diarrhea), assuming an event rate of 15% in the control group (2-tailed α = 0.05). We targeted enrolling 300 patients to allow some room for error in our assumptions. null hypothesis: incidence of diarrhea is no different between the aminophylline arm and the placebo arm; Test type: Superiority or Other; p = 0.002, Chi-squared

2. Secondary Outcome: Number of Patients With Any (One or More) Regadenoson-related Adverse-effect
Description: Regadenoson-related adverse-effects include: flushing, feeling hot, chest pain, chest discomfort, angina, headache, dizziness, abdominal cramps or discomfort, diarrhea, nausea.
  When multiple adverse effects are reported, only one event is counted.
Time Frame: Within 2 hours from the intervention.
Population: All patients.
Measure: Number; unit: Participants
Arm/Group | Aminophylline | Placebo
Number analyzed (Participants) | 150 | 150
Participants | 47 | 96
Statistical Analysis 1: Comparison: Aminophylline vs Placebo; Test type: Superiority or Other; p < 0.001, Chi-squared

3. Secondary Outcome: Global Symptom Score (GSS) of Regadenoson Related Adverse-effects
Description: GSS is the sum of severity-weighted (0 = none, 1 = mild, 2 = moderate, 3 = severe) regadenosnon-related adverse-effects of flushing, feeling hot, chest pain, chest discomfort, angina, headache, dizziness, abdominal cramps or discomfort, diarrhea, nausea.
  GSS is calculated by weighting each side effect from 0 - 3 (as above) then add the severity weighted scores of all adverse effects (total of 10 as above).
  The number of adverse effects contributing to the score is 10, each has a potential severity weight of 0 (absent) to 3 (severe). Thus:
  Minimum possible Global Symptom Score (GSS) = 0 Maximum possible Global Symptom Score (GSS) = 30
Time Frame: Within 2 hours from the intervention.
Population: All patients.
Measure: Mean (Standard Deviation); unit: Global Symptom Score
Arm/Group | Aminophylline | Placebo
Number analyzed (Participants) | 150 | 150
Global Symptom Score | 1.7 (0.8) | 2.1 (1.6)
Statistical Analysis 1: Comparison: Aminophylline vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Patients With Recorded Aminophylline Related Major Adverse Events
Description: Aminophylline related adverse effects include: systemic hypotension (systolic blood pressure < 90 mmHg), any thachyarrhythmia (ventricular or supraventricular) and seizure.
Time Frame: Within 24 hours from the intervention.
Population: All patients.
Measure: Number; unit: participant
Arm/Group | Aminophylline | Placebo
Number analyzed (Participants) | 150 | 150
participant | 0 | 0
Statistical Analysis 1: Comparison: Aminophylline vs Placebo; Test type: Superiority or Other; p = 1, Chi-squared

ADVERSE EVENTS:
Time Frame: 24 hours
Description: In addition to all-cause mortality, the following adverse effects (AEs) were monitored and reported:
  1. Tachyarrhythmias: any tachyarrhythmia within the subsequent 24 hours, not present baseline
  2. Hypotension: any event of systolic blood pressure =/< 80 mmHg regardless of symptoms or systolic blood pressure =/< 90 mmHg with symptoms (dizziness, lightheadedness, presyncope, or syncope)
  3. seizures: any seizure event reported within the 24 hours following the initiation of the stress protocol
Arm/Group | Aminophylline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/150
Other Adverse Events (participants affected / at risk) | 0/150 | 0/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aminophylline (N=150) | Placebo (N=150)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) — Tachyarrhythmia requiring treatment
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) — Systolic blood pressure equal or less than 80 mmHg
Seizure (Nervous system disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes